CLINICAL TRIAL: NCT00039507
Title: Pilot Study: Radiofrequency Ablation Of Resectable Non-Small Cell Lung Cancer
Brief Title: Radiofrequency Ablation During Surgery in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069389; P30CA006927 (NIH); FCCC-02007; NCI-G02-2079
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiofrequency Ablation

INTERVENTIONS:
Procedure: conventional surgery
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency ablation uses high-frequency electric current to kill tumor cells. Combining radiofrequency ablation with surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining radiofrequency ablation with surgery in treating patients who have stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the acute effects of intraoperative radiofrequency tumor ablation (RFA) in patients with resectable non-small cell lung cancer.
* Determine the treatment-related toxicity in patients treated with this therapy.
* Determine the dimensions of the RFA lesion produced by the ablation procedure in these patients.

OUTLINE: Patients undergo intraoperative radiofrequency tumor ablation over 10-15 minutes for each tumor immediately followed by tumor resection.

PROJECTED ACCRUAL: A maximum of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of malignant non-small cell lung cancer (NSCLC)

  * Intraoperative needle biopsy confirmation allowed
* Resectable disease (stage I or II)
* All tissue to be treated by radiofrequency tumor ablation must be completely contained within boundaries of planned lung resection
* Medically fit to undergo lung resection

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior or concurrent biologic therapy

Chemotherapy:

* No prior or concurrent chemotherapy

Endocrine therapy:

* No prior or concurrent endocrine therapy

Radiotherapy:

* No prior or concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No other prior therapy for NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter J. Scott, MD, FACS, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States